CLINICAL TRIAL: NCT04167592
Title: Effectivity of Benzydamine Hydrochloride Gargle to Reduce Propofol Consumption in Endoscopic Retrograde Cholangiopancreatography Procedure
Brief Title: Benzydamine Hydrochloride Gargle in Reducing Propofol for ERCP
Acronym: ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Adhrie Sugiarto, Medical Staff, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes041
Record Dates: First submitted 2019-11-08; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: ERCP
Keywords: propofol; benzydamine hydrochloride; sore throat; Endoscopic Retrograde Cholangiopancreatography
MeSH Terms: conditions — Pharyngitis | interventions — Benzydamine; Mouthwashes; Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benzydamine Hydrochloride Group (Active Comparator): Subjects who were allocated in benzydamine group would gargle with 15 of ml benzydamine hydrochloride 0.15% before sedation started.
  Interventions: Drug: Benzydamine Hydrochloride 0.15% Oral Rinse
- Control Group (Placebo Comparator): Subjects who were allocated in control group would gargle with 15 ml of water before sedation started.
  Interventions: Drug: Water

INTERVENTIONS:
Drug: Benzydamine Hydrochloride 0.15% Oral Rinse — Benzydamine Hydrochloride 0.15% Oral Rinse was used to gargle prior to Endoscopic Retrograde Cholangiopancreatography (ERCP) procedure.
  Arms: Benzydamine Hydrochloride Group
Drug: Water — Water was used to gargle prior to Endoscopic Retrograde Cholangiopancreatography (ERCP) procedure.
  Arms: Control Group

SUMMARY:
It was a study aimed to determine the effectivity of benzydamine hydrochloride gargling in reducing propofol consumption in the Endoscopic Retrograde Cholangiopancreatography (ERCP) procedure.

DETAILED DESCRIPTION:
The study was approved by Ethics Committee of Indonesia University. It was a single-blind randomized clinical trial at Cipto Mangunkusumo Hospital - Jakarta during August to September 2018. 72 subjects were recruited and randomly assigned into 2 groups. Patients in group B were given 0.15% mouthwash with benzydamine hydrochloride prior to procedure while patients in group C were given mouthwash with 15 ml of water. Cumulative propofol consumption per minute per kg body weight, and incidence of postoperative sore throat were measured for each group.

ELIGIBILITY:
Inclusion Criteria:

* undergoing ERCP
* ASA I-III
* BMI 18-30 kg/m2

Exclusion Criteria:

* allergic to propofol
* contraindicated to propofol
* had throat wound or laceration
* received analgesics or steroid in 24 hours priorly
* unstable during sedation
* procedure longer than 90 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Cumulative Propofol Consumption | 90 minutes
  About 1 mg/kg Propofol was initially administered to sedate the subjects. If the subject's RSS (Ramsay Sedation Scale) rose, 0.3 mg/kg was additionally given. The amount of propofol used, as in mg/kg, during the ERCP procedure was recorded.
Incidence of Sore Throat | 4 hours
  Sore throat incidence after ERCP procedure was recorded

CONTACTS AND LOCATIONS:
Overall Officials: Adhrie Sugiarto, MD, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Triantafillidis JK, Merikas E, Nikolakis D, Papalois AE. Sedation in gastrointestinal endoscopy: current issues. World J Gastroenterol. 2013 Jan 28;19(4):463-81. doi: 10.3748/wjg.v19.i4.463. PMID 23382625
- [Background] Yang JF, Farooq P, Zwilling K, Patel D, Siddiqui AA. Efficacy and Safety of Propofol-Mediated Sedation for Outpatient Endoscopic Retrograde Cholangiopancreatography (ERCP). Dig Dis Sci. 2016 Jun;61(6):1686-91. doi: 10.1007/s10620-016-4043-3. Epub 2016 Jan 29. PMID 26825844
- [Background] Kati I, Tekin M, Silay E, Huseyinoglu UA, Yildiz H. Does benzydamine hydrochloride applied preemptively reduce sore throat due to laryngeal mask airway? Anesth Analg. 2004 Sep;99(3):710-712. doi: 10.1213/01.ANE.0000133142.52961.8D. PMID 15333399
- [Derived] Sugiarto A, Kapuangan C, Tantri AR, Chrisnata V. Effectivity of benzydamine hydrochloride gargle to reduce propofol consumption in endoscopic retrograde cholangiopancreatography procedure: a randomized controlled trial. BMC Anesthesiol. 2020 May 23;20(1):123. doi: 10.1186/s12871-020-00996-x. PMID 32446304